CLINICAL TRIAL: NCT03069703
Title: Multicenter Randomized Controlled Trial Comparing Immunogenicity and Safety of Two Innovative Anti-pneumococcal Vaccine Strategies to Standard Vaccination Regimen in Patients With ANCA-associated Vasculitis Receiving Rituximab Therapy
Brief Title: Innovative Anti-pneumococcal Vaccine Strategies in Patients With ANCA-associated Vasculitis Receiving Rituximab Therapy
Acronym: PNEUMOVAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: EUCLID Clinical Trial Platform (Other); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); CIC 1417 Cochin-Pasteur (Other); Groupe Français d'Etude des Vascularites (GFEV) (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P150964; 2016-002888-33 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Invasive Pneumococcal Infection
Keywords: Vaccine; ANCA- associated vasculitides; pneumovax; prevenar; pneumovas
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines; Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The central laboratory performing the immunogenicity assessment (ELISA and OPA) will be blinded for the trial arm in order to limit measurement bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prime-boost strategy (Active Comparator): a single dose of 13-valent pneumococcal conjugate vaccine (Prevenar, PCV13) at Day 0 (lying within a window of ± 2 days of the first infusion of rituximab), followed by a single dose of 23-valent unconjugated vaccine (Pneumovax, PPV23) at month 5 (M5)
  Interventions: Biological: PCV13; Biological: PPV23; Drug: Rituximab
- Innovative vaccine strategy 1 (Experimental): 2 doses of PCV13 at Day 0 and 2 doses of PCV13 at Day 7, followed by a single dose of PPV23 at M5
  Interventions: Biological: PCV13; Biological: PPV23; Drug: Rituximab
- Innovative vaccine strategy 2 (Experimental): 4 doses of PCV13 at Day 0, followed by a single dose of PPV23 at M5
  Interventions: Biological: PCV13; Biological: PPV23; Drug: Rituximab

INTERVENTIONS:
Biological: PCV13 — one dose of PCV13 at D0 (arm A) or two double doses at D0 and D7 (Arm B) or one quadruple dose at D0 (arm C)
  Other Names: Prevenar
Biological: PPV23 — one dose of PPV23 at M5
  Other Names: Pneumovax
Drug: Rituximab — 375 mg/m2/week for 4 consecutive weeks, at Days 0 ± 2 days, Day 7 ± 2 days, Day 14 ± 2 days and Day 21 ± 2 days, as induction therapy of vasculitis flare, followed by 500 mg-rituximab infusion every 6 months as maintenance therapy, i.e. at Month 6, Month 12 and Month 18

SUMMARY:
The study hypothesis is that a "reinforced" pneumococcal combined vaccine strategy in patients with ANCA-associated vasculitides treated with rituximab will induce a better immune response than the current standard regimen, with an acceptable safety profile.

This study therefore aims at evaluating the immunogenicity and safety of two "reinforced" innovative pneumococcal vaccine regimen [one double dose at day0 and one double dose at day7 or a quadruple dose of 13-valent anti-pneumococcal conjugate vaccine (PCV13) followed by one dose of 23-valent unconjugated vaccine (PPV23) at month 5], compared to the standard regimen (one dose of PCV13 followed by one dose of PPV23 at month 5), in patients with ANCA-associated vasculitides receiving rituximab therapy.

DETAILED DESCRIPTION:
Description of research methodology

Experimental plan This is a comparative, multicenter, prospective, randomized, open label, phase 2 trial in France, comparing two innovative "reinforced" anti-pneumococcal vaccine strategies to standard vaccination regimen in patients with ANCA-associated vasculitides receiving rituximab therapy.

Participants will be randomized 1:1:1 to three parallel arms to receive:

* Arm A (standard vaccination regimen): prime-boost strategy combining a single dose of 13-valent pneumococcal conjugate vaccine (Prevenar, PCV13) at Day 0 (lying within a window of ± 2 days of the first infusion of rituximab), followed by a single dose of 23-valent unconjugated vaccine (Pneumovax, PPV23) at month 5 (M5)
* Arm B (innovative vaccine strategy 1): prime-boost strategy combining 2 doses of PCV13 at Day 0 and 2 doses of PCV13 at Day 7, followed by a single dose of PPV23 at M5
* Arm C (innovative vaccine strategy 2): prime-boost strategy combining 4 doses of PCV13 at Day 0, followed by a single dose of PPV23 at M5

All participants will receive rituximab at 375 mg/m2/week for 4 consecutive weeks, at Days 0 ± 2 days, Day 7 ± 2 days, Day 14 ± 2 days and Day 21 ± 2 days, as induction therapy of vasculitis flare, followed by 500 mg-rituximab infusion every 6 months as maintenance therapy, i.e. at Month 6, Month 12 and Month 18 (Stone, NEJM, 2010, Jones, NEJM, 2010; Guillevin, NEJM, 2014), as recommended.

Day 0 will be defined as the first vaccine injection (within ± 2 days of the first infusion of rituximab).

PCV13 vaccine injections will be performed at Day 0, and at Day 7 ± 1 day in the Arm B. PPV23 injections will be performed at M5 ± 7 days in all arms.

Analysis of immune responses will be performed in a centralized laboratory blinded for the trial arm, by ELISA at Day 0 (pre-vaccination sample), M1, M5, M6, M12, and M18 for the 12 serotypes common to both conjugate and unconjugated vaccines, by OPA at Day 0, M6, M12, and M18 for the 12 serotypes common to both conjugate and unconjugated vaccines, and by ELISA at Day 0 and M6 for the 3 specific serotypes of PPV23.

Safety monitoring Relevant adverse events related to vaccination will be continuously monitored throughout the trial, and pausing rules have been specified in the protocol that trigger an ad-hoc iDSMB meeting in case of any safety concern

Number of participating centres

This multicenter research will involve the participation of the French Vasculitis Study Group (FVSG) network, which includes more than 100 clinical departments involved in the management of ANCA-associated vasculitides.

As previous trials conducted by the FVSG on this topic, around 50 centers will participate in the PNEUMOVAS research.

Randomization Participants who fulfill all eligibility criteria for the study will be enrolled and randomized in a ratio of 1:1:1 between the three different parallel arms.

Randomization will be stratified on: personal history of PPV23 injection and age (≥ 65 or < 65 years).

Blinding methods and provisions put in place to maintain blinding

Trial participants and site staff are not blinded to the vaccine arm. The central laboratory performing the immunogenicity assessment (ELISA and OPA) will be blinded for the trial arm in order to limit measurement bias.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a diagnosis of ANCA-associated vasculitis, either granulomatosis with polyangiitis (GPA, Wegener) or microscopic polyangiitis (MPA), according to ACR 1990 criteria and/or revised Chapel Hill Consensus Conference definitions and/or European Medical Agency algorithm
2. Participants (males and females) aged of 18 years or older
3. Participants with childbearing potential having reliable contraception for all the duration of the study, such as established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) or true abstinence (when this is in line with the preferred and usual lifestyle of the subject) prior to enrollment at D0
4. Participants with newly-diagnosed disease at the time of inclusion or presenting with a relapse of the disease. For relapsing patients, maintenance therapy at stable dose during the last 3 months will be admitted : prednisone dose ≤10 mg/day, azathioprine dose ≤3 mg/kg/day, methotrexate dose ≤25 mg/week, or mycophenolate mofetil dose ≤3 g/j
5. Participants with an active disease defined as a BVAS ≥ 3
6. Participants planned to receive rituximab as induction therapy using the recommended regimen (i.e. 375 mg/m2/week for 4 consecutive weeks)
7. Participants able to give written informed consent prior to participation in the study
8. Participants covered by social security regimen or equivalent

Exclusion Criteria:

1. Participants with eosinophilic granulomatosis with polyangiitis (EGPA, Churg-Strauss) or other vasculitis
2. Participants with acute infections or chronic active infections at inclusion visit.
3. Documented positive serology result for HIV, HBV (Ag Hbs), HCV at inclusion.
4. Participants with disease associated with decreased immune response (splenectomy, hematopoietic stem cell transplantation, primary immune deficiency such as common variable immunodeficiency, cancer within the previous 5 years, drepanocytosis),
5. Participants treated with rituximab within the previous 12 months,
6. Participants who have received blood, blood products, and/or plasma derivatives including parenteral immunoglobulin preparations in the past 3 months before enrolment.
7. Participants treated with new other immunosuppressive or immunomodulatory agents within the previous 3 months (including cyclophosphamide, anti-TNF-alpha, intravenous immunoglobulins, abatacept),
8. Participants treated with prednisone dose >10 mg/day for a duration greater than 21 days before inclusion,
9. Participants with vaccination with a conjugate anti-pneumococcal vaccine at any time,
10. Participants with vaccination with PPV23 within the previous 3 years,
11. . Participants who have received any another vaccines within 4 weeks prior to enrolment or who are planning to receive any vaccine within the first 6 months of the study (except annual influenza vaccination and hepatitis B virus vaccination which are permitted before and after each vaccination visit of the study and then allowed at any time during the study follow up).
12. Pregnant women and lactation,
13. Participants with contraindication to use rituximab,
14. Participants with contraindication to intramuscular injections (hemophilia, anticoagulant therapy (excepted if subcutaneously), thrombocytopenia < 50 000/mm3).
15. Participants with hypersensitivity to previous vaccination
16. Participants with hypersensitivity to aluminium phosphate, phenol or protein CRM197 protein from Corynebacterium diphtheria.
17. Participants included in another investigational therapeutic study in the month prior D0. Participation to an observational research is allowed.
18. Participants under legal guardianship or incapacitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 6 months
  Immune response at M6 against 12 pneumococcal serotypes, according to four ordered categories of response: positive response to 0-3, 4-6, 7-9, or 10-12 serotypes common to the PCV13 and PPV23 vaccines. This endpoint will be analyzed as the number and proportion of participants in each of the four response categories using a proportional odds model

SECONDARY OUTCOMES:
Local and/or systemic solicited reactions 7 days following each vaccination | 18 months
  proportion of participants with an event; number, nature, grade and time of occurrence.
Any adverse event during the trial related or possibly related to vaccine immunization | 18 months
  proportion of participants with an event; number, nature, grade and time of occurrence.

OTHER OUTCOMES:
Any adverse event during the trial related to vaccine immunization and leading to discontinuation of the immunization regimen | 18 months
  proportion of participants with an event; number, nature, grade and time of occurrence;
Any serious adverse event during the study, regardless of the relationship to vaccine immunisation | 18 months
  proportion, number, nature, grade and time of occurrence
Proportion of patients with vasculitis flare according to EULAR criteria during the study period, and time to disease relapse. | 18 months
Titer of specific IgG against the 12 serotypes common to both conjugate and unconjugated vaccines (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F) measured by OPA at Day 0 and M6 | 6 months
Titer of specific IgG against the 3 specific serotypes of PPV23 (10A, 12F et 15B) at Day 0 and M6 | 6 months
Titer of specific IgG against the 12 serotypes common to both conjugate and unconjugated vaccines (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F) measured by ELISA at M1 and M5 | 5 months
Titer of specific IgG against the 12 serotypes common to both conjugate and unconjugated vaccines (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F) measured by ELISA at M12 and M18 | 18 months
Titer of specific IgG against the 12 serotypes common to both conjugate and unconjugated vaccines (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19 A, 19F and 23F) measured by OPA at M12 and M18 | 18 months
Frequency of occurrence of invasive pneumococcal infections in the different vaccine strategies | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin TERRIER, MD, PhD, Principal Investigator — Pôle de Médecine Interne, Centre de référence " Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques " Hôpital Cochin, Assistance Publique-Hôpitaux de Paris; Fréderic BATTEUX, PhD, Study Chair — Laboratoire d'Immunologie Plateforme d'immunomonitoring vaccinal Hôpital Cochin, Assistance Publique-Hôpitaux de Paris; Odile LAUNAY, MD, PhD, Principal Investigator — Centre d'Investigation Clinique Cochin Pasteur Hôpital Cochin, Assistance Publique-Hôpitaux de Paris; Matthieu GROH, MD, Principal Investigator — Hôpital Foch
Locations (1):
- Pôle de Médecine Interne, Centre de référence " Maladies systémiques et autoimmunes rares, en particulier Vascularites nécrosantes et Sclérodermies systémiques " Hôpital Cochin, Assistance Publique-Hôpitaux de Paris, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] doi:10.1136/ard.2010.137778
- [Background] doi:10.1136/ard.2008.088302
- [Background] Nazi I, Kelton JG, Larche M, Snider DP, Heddle NM, Crowther MA, Cook RJ, Tinmouth AT, Mangel J, Arnold DM. The effect of rituximab on vaccine responses in patients with immune thrombocytopenia. Blood. 2013 Sep 12;122(11):1946-53. doi: 10.1182/blood-2013-04-494096. Epub 2013 Jul 12. PMID 23851398
- [Background] doi:10.1016/j.vaccine.2011.04.132
- [Background] McGregor JG, Negrete-Lopez R, Poulton CJ, Kidd JM, Katsanos SL, Goetz L, Hu Y, Nachman PH, Falk RJ, Hogan SL. Adverse events and infectious burden, microbes and temporal outline from immunosuppressive therapy in antineutrophil cytoplasmic antibody-associated vasculitis with native renal function. Nephrol Dial Transplant. 2015 Apr;30 Suppl 1(Suppl 1):i171-81. doi: 10.1093/ndt/gfv045. PMID 25805747
- See also: Website of the necrotizing vasculitides reference center — http://www.vascularites.org/
- See also: Website of the vaccinology clinical center Pasteur Cochin — http://www.cicvaccinologie.com/